CLINICAL TRIAL: NCT04101682
Title: Continuous Vs Single Shot Adductor Canal Block After ACL Reconstruction - A Randomized Study
Brief Title: Continuous Vs Single Shot Block After ACL
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not enough enrollment
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0811
Record Dates: First submitted 2019-08-26; First posted 2019-09-24 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Shot (Active Comparator): Patients will receive an adductor canal block in the operating room postoperatively as single shot of 20-30cc bupivacaine
  Interventions: Drug: Bupivacaine
- Continuous Block (Active Comparator): Patients will have a catheter inserted into the adductor canal which will be attached up to a continuous infusion pump of bupivacaine that will have a set flow rate over the next couple days
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Administered by an anesthesiologist or certified nurse anesthetist, under ultrasound guidance a catheter placed overlying the nerve sheath. This catheter is then connected to a device with a reservoir that administers local anesthetic at a set rate.

SUMMARY:
The investigators will be randomizing patients to either receive an adductor canal block in the operating room postoperatively as single shot of 20-30cc bupivacaine or to have a catheter inserted into the adductor canal which will be attached up to a continuous infusion pump of bupivacaine that will have a set flow rate over the next couple days. The investigators' hypothesis is that patients will have better pain control, sleep, and decreased opioid consumption with the use of a continuous infusion pump

DETAILED DESCRIPTION:
Screening evaluation will occur during the preoperative visit prior to surgery which generally occurs within 28 days prior to surgery. No separate screening is indicated in this study.

Patients will be asked to participate in the study if they are having ACL Reconstruction surgery with one of the orthopedic surgeons who is participating in the study. They will be informed and consented in the office or in the preoperative holding area prior to surgery.

Patients undergo ACL reconstruction at either Plainview, Franklin, Huntington, Long Island Jewish, or North Shore University Hospital.

Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an adverse event (AE). However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

The investigator who is making phone calls to the given participant will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit/phone call, the investigator will inquire about the occurrence of AE/SAEs since the last visit/phone call. Events will be followed for outcome information until resolution or stabilization.

Study procedures and evaluations

* All patients who are enrolled in this study will have been evaluated and determined to be a candidate for ACL reconstruction surgery. The indications for surgery, determination of need for surgery and physical examination determining this need are independent from the interventions and outcomes being assessed by this study.
* Efficacy Assessment plan- All patients will be called on postoperative days 1,2,3,4, 7 via and be assessed in person at the post-operative visit. They will be surveyed for primary and secondary outcomes by a study investigator. Primary outcome will be assessed using visual analog scale 0-10. Secondary outcomes; Opiate consumption will be assessed documented during the phone call, Sleep will be assessed by either yes or no answer if the patient had a disturbance in their sleep or had trouble getting to sleep based on pain of the surgical knee in the past 24 hours.
* Screening evaluation will occur during the preoperative visit prior to surgery which generally occurs within 28 days prior to surgery. No separate screening is indicated in this study.
* Procedure for administering study intervention and follow-up procedures. The participant will be seen in the preoperative holding suite prior to surgery to ensure that patient is still willing to undergo randomization for the study. The patient will then undergo randomization by a computer-based software and the anesthesiologist will be informed of the plan. The participant will undergo anesthesia at the discretion of the anesthesiologist per routine given the participant's clinical baseline. The participant will undergo ACL reconstruction based on the standard of care treatment. Following surgery but prior to leaving the operating room the anesthesiologist will place the adductor canal block and the catheter based on the participant's randomization under ultrasound guidance to ensure proper placement of the block. The participant will then undergo routine post-operative care in the recovery suite with routine recovery room vital checks. For participants who are randomized to the continuous pump group, the pump will be assembled and filled by pharmacy and attached to the previously placed catheter while the participant is in the recovery room. Once the participants are awake and alert in the recovery room, a study investigator will review the study specifics again, including the phone calls with written information on the questions that will be asked. They will also be given written instructions on how to use the continuous pumps and how to remove it. If the patient is uncomfortable removing it themselves, they can come to the office to have it removed. For participants who received a continuous pump the investigator will go over the function of the pump, troubleshooting, and how to remove the pump at home. All participants will be discharged home from the recovery room after they have met the routine discharge criteria following existing standard of care recovery room protocols.
* All data will be recorded in an encrypted database which is HIPPA and IRB compliant. All participant information will be labeled with a participant study identification number with no identifiable information documented.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged >16 years old
* In good general health as evidenced by medical history and deemed medically healthy enough to tolerate surgery by the patient's primary care physician
* MRI with evidence of ACL tear, and wanting to have an ACL reconstruction surgery
* Ability to take oral medication and be willing to adhere to the study intervention, including telephone calls
* Agrees to complete surveys required on the days specified between 5-9PM

Exclusion Criteria:

* Current daily opioid requirement exceeding the equivalent of 15mg morphine
* Daily prescription of corticosteroid, tricyclic antidepressant, gabapentin, or tramadol
* Carrying the diagnosis of chronic pain syndrome, uncontrolled anxiety, history of schizophrenia or related psychiatric disorders
* History of alcohol or drug abuse/addiction
* History of preexisting nerve damage in the surgical extremity
* Knee surgery (same knee) in the previous 12 weeks
* Anticipated knee surgery in the other knee planned in the ensuing 6 months
* Diabetic patients with blood sugar values exceeding 250 mg/dl in the previous month
* BMI >40Kg/m2
* Pregnancy, which will be determined by a serum or urine HCG test on the day of surgery.
* Incarceration
* Inability to communicate with staff, including being unreachable by telephone
* Revision ACL reconstruction
* Patient reconsideration after initial agreement.
* Non-English speaking subjects

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Pain at Rest | Day 1
  Measured by a visual analogue scale (1-10)
Pain at Rest | Day 2
  Measured by a visual analogue scale (1-10)
Pain at Rest | Day 3
  Measured by a visual analogue scale (1-10)
Pain at Rest | Day 4
  Measured by a visual analogue scale (1-10)
Pain at Rest | Day 7
  Measured by a visual analogue scale (1-10)
Pain at Rest | Day 14
  Measured by a visual analogue scale (1-10)
Worst Pain in the past 24 hours | Day 1
  Measured by visual analogue scale 1-10
Worst Pain in the past 24 hours | Day 2
  Measured by visual analogue scale 1-10
Worst Pain in the past 24 hours | Day 3
  Measured by visual analogue scale 1-10
Worst Pain in the past 24 hours | Day 4
  Measured by visual analogue scale 1-10
Worst Pain in the past 24 hours | Day 7
  Measured by visual analogue scale 1-10
Worst Pain in the past 24 hours | Day 14
  Measured by visual analogue scale 1-10

SECONDARY OUTCOMES:
Daily Opioid Consumption | on post operative day 1,2,3,4,7, and 14
  This will be measured as daily consumption of oxycodone (morphine equivalents)
Incidence of Disturbed Sleep | on post operative day 1,2,3,4,7, and day 14
  Measured this by asking if they had a disturbance in their sleep or trouble getting to sleep because of pain in the surgical knee
IKDC - International Knee Documentation Commitee Form for Knee Function | Preoperatively, 3 months, 6 months
  Subjective validated scoring form for knee function. Scale 0-10. 0 for not being able to perform any function. 10 being no limitation in function
Rand Short Form - 36 | Preoperatively, 3 months, 6 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health

CONTACTS AND LOCATIONS:
Overall Officials: Randy Cohn, MD, Principal Investigator — Northwell Health
Locations (1):
- Plainview Hospital, Plainview, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT04101682/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT04101682/ICF_001.pdf